CLINICAL TRIAL: NCT03539315
Title: Adaptation and Testing of the Addressing Reproductive Coercion in HEalth Settings (ARCHES) Intervention to Improve Reproductive Autonomy and Reproductive Health Among Abortion Clients in Bangladesh
Brief Title: Adaptation and Testing of the Addressing Reproductive Coercion in HEalth Settings (ARCHES) Intervention in Bangladesh
Acronym: ARCHES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ipas (Other)
Collaborators: University of California, San Diego (Other); Ipas Bangladesh (Unknown); Bangladesh Association for Prevention of Septic Abortion (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BD_01
Record Dates: First submitted 2018-05-14; First posted 2018-05-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2020-02

CONDITIONS: Violence, Domestic
MeSH Terms: interventions — cpsf4 protein, zebrafish

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: ARCHES (Experimental): All women attending facilities assigned to the intervention arm receive the Addressing Reproductive Coercion within Healthcare Settings (ARCHES) intervention.
  Interventions: Behavioral: ARCHES
- Control (No Intervention): All women attending facilities assigned to the control arm receive the standard of care (no intervention).

INTERVENTIONS:
Behavioral: ARCHES — Addressing Reproductive Coercion within Healthcare Settings (ARCHES) is a clinic-based intervention developed in the U.S., and involves training existing health providers to identify RC and IPV during standard family planning clinic-based counselling interactions. The intervention seeks to empower women with harm reduction strategies that minimize their risk for unintended pregnancy by offering a wide range of contraceptive options, providing counseling on correct and consistent use of contraception, and counseling on contraceptive methods that are difficult for a male partner to detect or block such as injectables or IUDs. ARCHES also facilitates access to violence support and counselling services by connecting women with community-based IPV services.
  Arms: Intervention: ARCHES

SUMMARY:
The primary purpose of this research is to conduct a brief project to adapt and evaluate an evidence-based intervention model to address reproductive coercion and unintended pregnancy (ARCHES - Addressing Reproductive Coercion within Healthcare Settings) to the Bangladesh cultural context and for use with abortion clients (i.e., develop ARCHES Bangladesh) so as to provide initial assessment of acceptability, feasibility and effectiveness in this high-need LMIC context. Globally, addressing violence and coercion from male partners is considered key to reducing unintended pregnancy among adult and adolescent women. This has led to multiple efforts to integrate IPV screening and counseling in health settings, particularly in the context of family planning, across a range of middle and low-income countries. However, to date, no existing model addressing reproductive coercion has demonstrated reduction in risk for unintended pregnancy, either for Bangladesh or any other country.

DETAILED DESCRIPTION:
Reproductive coercion and partner violence are associated with unwanted pregnancy and abortion globally. In Bangladesh, women reporting partner violence are more likely to access abortion outside the health system and less likely to access post-abortion contraception, especially if accompanied to the clinic by their partner, which suggests additional intervention is needed to support clients' reproductive autonomy and ultimately their ability to safely control their fertility. ARCHES (Addressing Reproductive Coercion in HEalth Settings) is a clinic-based harm reduction intervention that empowers women to implement strategies that mitigate the impact of reproductive coercion on their reproductive health. ARCHES has been shown to reduce reproductive coercion among family planning clients in the U.S., but it has not previously been used in Asia or specifically with MR/PAC clients. This study seeks to adapt the ARCHES intervention for use with MR/PAC clients in Bangladesh and to test its effectiveness through a cluster randomized controlled trial. Overall, this study is expected to result in 1) evidence of the effectiveness of the adapted ARCHES intervention in increasing contraceptive use and reducing reproductive coercion, and ultimately in reducing the risk for future unintended pregnancy and unsafe abortion, and 2) evidence on the elements required for successful implementation in high volume MR/PAC clinics.

The aims of this study are:

1. To conduct formative work to inform the adaptation of the ARCHES intervention to the Bangladesh context and for use with abortion clients.
2. To pilot the adapted intervention
3. To test the effect of the adapted ARCHES intervention on uninterrupted contraceptive use and reproductive coercion, and ultimately reduction in future unintended pregnancy and unsafe abortion, among abortion clients in Bangladesh.
4. To evaluate implementation of the ARCHES intervention using an implementation science approach.
5. To understand out of clinic abortion attempts and how these attempts interact with women's experiences of violence.
6. To assess structural, community-related, and cultural barriers to accessing MR, methods of self-induced abortion, and abortion care received prior to presenting for MR/PAC.

ELIGIBILITY:
Inclusion Criteria:

* Woman receiving MR or PAC services during the evaluation phase in all 6 selected RHSTEP clinics
* Age 18-49
* Able to provide a safe phone number at which they can be contacted for study follow-up
* Not being accompanied to the clinic by a person (e.g. spouse, family member) who refuses to allow her to be spoken to privately by the provider and/or research assistant
* Able to provide informed consent
* Able to communicate in Bangla
* Not planning on moving out of the area in the coming year

Exclusion Criteria:

* Woman not receiving MR or PAC services during the evaluation phase in the 6 selected RHSTEP clinics
* Not age 18-49
* Unable to provide a safe phone number for follow-up
* Accompanied to the clinic by a person (e.g. spouse, family member) who refuses to allow her to be spoken to privately by the provider and/or research assistant
* Unable to provide informed consent
* Unable to communicate in Bangla
* Planning on moving out of the area in the coming year

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Woman receiving abortion services
Enrollment: 2729 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Modern contraceptive use without interruption or partner interference | Past 4 months
  Proportion of women reporting use of a modern contraceptive method (pills, condoms, injectables, IUD, implant, sterilization) without reported interruption or partner interference such as contraceptive sabotage.

SECONDARY OUTCOMES:
Reproductive coercion | Past 4 months
  Proportion of women reporting reproductive coercion. A reproductive coercion metric for Bangladesh is currently under development. Reproductive coercion metrics used in other settings include indicators such as contraceptive sabotage, a husband or family member preventing a woman from accessing contraception, and pressure for her to become pregnant when she does not wish to be pregnant. This description will be replaced with the reproductive coercion metric developed for Bangladesh when it is available.
Unsafe abortion | Past 12 months
  Proportion of women reporting accessing unsafe abortion services, including an unsafe provider (provider who is untrained or unauthorized to provide abortion services) or using an unsafe method of abortion (a method that is not a WHO-approved uterine evacuation method).
Unintended pregnancy | Past 12 months
  Proportion of women reporting that when they got pregnant, they did not want to get pregnant at that time.

CONTACTS AND LOCATIONS:
Overall Officials: Erin E Pearson, PhD, Principal Investigator — Ipas
Locations (6):
- Bangladesh (6):
  - Chittagong Medical College Hospital RHSTEP Clinic, Chittagong
  - Dhaka Medical College Hospital RHSTEP Clinic, Dhaka
  - Faridpur Medical College Hospital RHSTEP Clinic, Farīdpur
  - Rajshahi Medical College Hospital RHSTEP Clinic, Rajshahi
  - Rangpur Medical College Hospital RHSTEP Clinic, Rangpur City
  - Sylhet Osmani Medical College Hospital RHSTEP Clinic, Sylhet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pearson E, Paul D, Menzel J, Shakhider MAH, Konika RA, Uysal J, Silverman JG. Effectiveness of the Addressing Reproductive Coercion in Health Settings (ARCHES) intervention among abortion clients in Bangladesh: a cluster-randomized controlled trial. EClinicalMedicine. 2024 Jun 28;73:102699. doi: 10.1016/j.eclinm.2024.102699. eCollection 2024 Jul. PMID 39040882